CLINICAL TRIAL: NCT06160388
Title: The Short- and Long-Term Safety of S53P4 Bioactive Glass for Mastoid Obliteration: a Retrospective Comparative Study
Brief Title: The Safety of S53P4 Bioactive Glass for Mastoid Obliteration
Status: Completed | Type: Observational
Sponsor: Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: 16-004-3
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Mastoid Cavity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients that underwent mastoidectomy + mastoid obliteration using bioactive glass: This is the intervention group, consisting of patients that have underwent either canal wall up or canal wall down mastoidectomy followed by obliteration of the mastoid cavity using S53P4 bioactive glass for any indication
  Interventions: Device: S53P4 Bioactive glass
- Patients that underwent mastoidectomy alone: This is the control group, consisting of patients that have underwent either canal wall up or canal wall down mastoidectomy without mastoid obliteration for any indication

INTERVENTIONS:
Device: S53P4 Bioactive glass — Following mastoidectomy, the mastoid cavity, and if the ossicular chain has been removed the epitympanum as well, are obliterated using S53P4 bioactive glass. The bioactive glass is mixed with saline and administered to the cavity, ensuring a tight fit.
  Groups: Patients that underwent mastoidectomy + mastoid obliteration using bioactive glass

SUMMARY:
In recent years, mastoid obliteration (MO) after mastoidectomy has gained popularity. However, the choice for obliteration material has been a point of discussion. Autologous materials have the advantage of being freely available without cost.Synthetic materials on the other hand have unlimited supply, hold volume over time and have no risk of donor site morbidity. Comparative studies between materials are rare and the few available were unable to ascertain superiority.

Our hospital has been utilizing the same material for obliteration since 2011: S53P4 bioactive glass (BAG). It since has become our main operating procedure to obliterate the mastoid cavity with BAG granules following both canal wall up (CWU) and canal wall down (CWD) mastoidectomy. This bioactive glass has several important characteristics, such as the retaining of volume over time and antibacterial properties.

An important factor when selecting obliteration material is safety. Data on this was reported in several studies, but unfortunately these studies only investigated short-term safety in small and selected cohorts of patients, often without comparison. Additionally, large studies with extensive follow-up are necessary to detect rare complications and long-term pitfalls. Therefore, the aim of this study is to determine the safety of BAG in a cohort that encompasses all cases that underwent CWU+MO and CWD+MO in our institute and compare these results to a non-obliteration cohort. The main outcomes are short- and long-term safety, as indicated by surgical complications in the first year following surgery and revision surgeries during follow-up, respectively. The investigators will compare the obliteration cohort to the non-obliteration cohort, hypothesizing that obliteration results in a comparable or lower rate of complications and revision surgeries

ELIGIBILITY:
Inclusion Criteria:

* Canal wall up or canal wall down mastoidectomy
* Operated between 2010 and 2022
* All indications are included

Exclusion Criteria:

* Other surgical techniques, such as subtotal petrosectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that were operated in our hospital using a canal wall up or canal wall down mastoidectomy between 2010 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1196 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with postoperative surgical complications in the first year following surgery | First year following surgery
  Complications that occured within the first year following surgery
  We compare the obliteration cohort to the non-obliterative cohort
The number of patients which require revision surgery during follow-up | At 3-, 5- and 8-years postoperatively
  Revision surgeries performed during follow-up due to problems with the obliteration

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Quak, MD, PhD, Principal Investigator — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided